CLINICAL TRIAL: NCT06199765
Title: Predictors of Perception on Risk of Needlestick Injury and Effectiveness of The Needlestick Prevention Module Among House Officers in Kelantan
Brief Title: Risk Perception of Needlestick Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Ahmed Farrasyah Bin Mohd Kutubudin, Doctor, Hospital Universiti Sains Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NMRR ID-23-00281-VRX
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Needlestick Injuries
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Intervention Model Description: All house officers who were eligible and consented, who participated in cross sectional study were included into intervention group until the required sample size was achieved. The same numbers of officers, eligible and consented were included into control group. For intervention, only educational intervention will be given which consist of lecture, demonstration, and role play. After that, data collection will be given right after the intervention completion and 4 weeks after that using self administered questionnaire. The same will be applied to the control group which data collection will be done right masking and 4 weeks later.
Who Masked: Participant
Masking Description: Control group will be given materials regarding patient safety as masking. Patient safety will have some element on needlestick and injury prevention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lecture, demonstration, and role play on NSI (Experimental): this arm will receive intervention regarding needlestick prevention using needlestick prevention educational module. this intervention only involve educational intervention which consist of lecture, demonstration, and role play. This intervention will be done for 1 week duration.
  Interventions: Other: Needlestick Injury Prevention
- Patient Safety Materials (Sham Comparator): This arm will receive material regarding patient safety. this material will have some element of needlestick and injury prevention. this intervention will done for 1 week.
  Interventions: Other: Needlestick Injury Prevention

INTERVENTIONS:
Other: Needlestick Injury Prevention — this intervention will be using needlestick injury prevention module which will involve lecture, demonstration, and role play

SUMMARY:
The purpose of this study is to determine the effectiveness of needlestick injury prevention module

DETAILED DESCRIPTION:
After being informed about the study and the potential risk, participants were given written informed consent to be filled out and signed. Agreed participants will receive a 1-week duration of educational intervention. The intervention only involved education and was less likely to cause injury or damage to the body.

ELIGIBILITY:
Inclusion Criteria:

1. All house officer in government hospitals with house officer training programme
2. House officers must be among those who join housemanship program for minimum of 1 month duration

Exclusion Criteria:

1. House officer who undergo attachment outside the training hospital
2. House officer that are not available during the data collection period or on long leave

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-19 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2024-01-11 (Estimated)

PRIMARY OUTCOMES:
Needlestick injury Risk Perception Score | right after intervention and 4 weeks after
  determine the risk perception score improvement using likert scale. 1 is the lowest and 5 is the highest mark. the higher the mark the better.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No